CLINICAL TRIAL: NCT04449367
Title: THE EFFECTIVENESS OF AN ULTRASOUND GUIDED RECTOR SPINAE BLOCK IN PATIENTS UNDERGOING THORACIC SPINE SURGERY
Brief Title: ERECTOR SPINAE BLOCK AFTER THORACIC SPINE SURGERY
Acronym: SPINE
Status: Completed | Type: Observational
Sponsor: Dubai Health Authority (Other Government)
Responsible Party: Principal Investigator, Dr Manar Mamdouh Fahmy Elsharkawi, SPECIALIST ANAESTHESIOLOGIST, Dubai Health Authority
Other Study IDs: DSREC-04/2018_01
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Post Operative Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Randomized and Single-Arm Trials: a sham comparator (no intervention)
  Interventions: Procedure: ultrasound guided erector spinae plane block

INTERVENTIONS:
Procedure: ultrasound guided erector spinae plane block — bilatral block given to patients under general anaesthesia for thoracic spine sugery to contorl post operative pain

SUMMARY:
the effectiveness of ultrasound guided erector spinae plane block in patients undergoing thoracic spine sugery

DETAILED DESCRIPTION:
bilateral erector spinae plane block would be given to patients with thoracic spine sugery for postoperative analgesia & its effectiveness would be evaluated for 2 days

ELIGIBILITY:
Inclusion Criteria:

* postoperative thoracic spine sugery

Exclusion Criteria:

* less then 18 years
* more than 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients underging thoracic spine sugery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-08-26 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
ultrasound guided erector spinae plane block can be used for postoperative analgesia for patients undergoing thoracic spine sugery | 2 days
  postoperative analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Dubai Health Authority, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No